CLINICAL TRIAL: NCT06933862
Title: Effects of Channa Striata Extract on Intestinal Inflammation and Nutritional Status in Malnutritional Toddlers After Albendazole Therapy in South Bangka District
Acronym: Striatin1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: Dexa Medica Group (Industry)
Responsible Party: Principal Investigator, Monica Puspa Sari, Head of Laboratory, Principal investigator, Fakultas Kedokteran Universitas Indonesia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MPuspaSari
Record Dates: First submitted 2025-03-12; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Malnourished Children
Keywords: snakehead fish extract; malnourished children; Calprotectin; striatin

STUDY DESIGN:
Intervention Model Description: The study participants were divided into 2 groups namely group A which received snakehead fish extract or inbumin forte sachet and group B which received a placebo. The study was conducted randomly and double blinded.
Who Masked: Participant, Investigator
Masking Description: Placebo controlled, Plasebo was made by PT Dexa Medica and randomization code was held by PT Dexa Medica.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Malnourished: Striatin (Experimental): Striatin or inbumin forte is given in the form of a 5 g dose of powder and 250 mg of curmicin. Striation or inbumin forte powder dissolved in 30 ml of drinking water and given one sachet per day, taken in the morning and evening after meals and given for 90 days
  Interventions: Dietary Supplement: Striatin
- Malnourished: Placebo (Placebo Comparator): placebo of striatin containing 4.89 g of mannitol was given in powder form and dissolved in 30 ml of drinking water. Placebo of striatin was given one sachet per day, taken in the morning and evening after meals and given for 90 days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Striatin — striation or placebo given for 90 days assigned to striatin
  Arms: Malnourished: Striatin
Dietary Supplement: Placebo — placebo
  Arms: Malnourished: Placebo

SUMMARY:
The goal of this clinical trial is to learn if intervention with channa striata extract or inbumin forte sachet as a food supplement can improve intestinal damage and nutritional status in malnourished children aged 1.5-5 years. The main questions it aims to answer are:

* Whether there is a change in calprotectin and AAT levels after administration of snakehead fish extract of inbumin forte sachet?
* Whether there is a difference in changes in nutritional status after administration of snakehead fish extract or inbumin forte sachet? Researchers will compare snakehead fish extract or inbumin forte sachet to a placebo (a look-alike substance that contains no drug) to see if snakehead fish extract or inbumin forte sachet works to treat children malnutrition.

Participants will take snakehead fish extract or inbumin forte sachet or placebo every day for 3 months. Researchers will visit study participants every month to check their weight and height and monitor vitamin administration through photos, notes and videos sent every day and records complaints or symptoms that may arise and at the end of 3 months, researchers will collect stool and blood samples and check nutritional status.

DETAILED DESCRIPTION:
The study participants were malnourished children aged 1.5 to 5 years. Data on malnourished children were obtained from the local health department. Based on this data, participants were selected from several sub-districts with the highest malnutrition cases, including Toboali (Rias and Toboali villages), Payung, Air Gegas, and Batu Betumpang sub-districts. After invitations were sent to the participants, they were registered using their family registration card and assigned a queue number or research code. The study plan and research procedures were then explained to the participants. First, anthropometric measurements were conducted including weight and height, with the results entered into the WHO Anthro calculator (-3 SD to <-2 SD). Baseline blood samples were collected, and labeled stool sample bottles were distributed. Fresh stool samples were collected the next day at a designated location. A 100 mg portion of each stool sample was transferred into a 1.5 ml Eppendorf tube and stored in a -20°C freezer. Each sample was divided into two tubes: one for gut microbiota analysis and the other for AAT and calprotectin testing using ELISA. Additionally, the Kato-Katz method was used to examine fresh stool samples for helminth infections. Following stool sample collection, participants were given albendazole at the appropriate dosage. Blood sample analysis included a complete blood count, amino acid testing using filter paper, serum ferritin using mini Vidas immunology analyzer, serum iron, total iron-binding capacity (TIBC) using Vitros chemistry analyzer and serum retinol levels using ELISA. Two weeks after albendazole administration, stool samples were re-examined using Kato-Katz method to confirm the absence of helminth infection. Then, participants were randomly assigned in a double-blind manner into two groups: one receiving snakehead fish extract (Inbumin Forte) and the other receiving a placebo. Based on sample size calculations, a minimum of 98 participants was required, and accounting for a 20% dropout rate, the total sample size was set at 122 children. Data processing was conducted using SPSS. A univariate analysis was performed to determine data distribution on ratio, nominal, and ordinal scales. Categorical data (nominal and ordinal) were presented as frequencies and percentages. Normality tests for numerical data were conducted using the Kolmogorov-Smirnov test, with a normal distribution determined if p > 0.05. Normally distributed data were presented as mean and standard deviation, while non-normally distributed data were shown as median and range (minimum-maximum).

Bivariate analysis was conducted to determine whether there were significant differences in nutritional status, macronutrient and micronutrient levels, inflammatory markers, intestinal permeability, and gut microbiota between children receiving striatin protein supplementation and those receiving a placebo. A paired t-test was used if the data were normally distributed to analyze mean differences between the two groups. If the data were not normally distributed, a chi-square test or Mann-Whitney test was applied. The effect of striatin protein intake on the studied variables was assessed using linear regression analysis. The hypothesis test results were interpreted at a 95% confidence level (α = 0.05), with the null hypothesis (H₀) being rejected if p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Malnourished children aged 1.5-5 years (-3SD to < -2 SD)
* Parents or guardians are willing to participate in the study
* Parents or guardians can read and fill out the questionnaire

Exclusion Criteria:

* Children with chronic diseases such as tuberculosis, congenital heart disease, diabetes, cancer, epilepsy, HIV Aids, sickle cell anemia, and mental illness.
* Children with history of snakehead fish allergy
* Children with physical disabilities that complicate data collection

Ages: 17 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 122 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Z-score (weight for age) | three months after intervention
  Z-score according to WHO antropometry that will be collected is based on weight for age. Body Weight in kg will be measured using a SECA brand weight scale. The differences between placebo and Inbumin Forte will be analysed after 3 months of treatment.
z-score (height for age) | three months after intervention
  Z-score according to WHO antropometry that will be collected is based on height for age. Height in cm will be using SECA brand height scale. The differences between placebo and Inbumin Forte will be analysed after 3 months of treatment.

SECONDARY OUTCOMES:
Concentrations of fecal calprotectin | From enrollment to the end of treatment at 3 months
  Calprotectin in stool samples were examined using ELISA (in mcg/g). The differences between placebo and Inbumin will be analysed at the end of 3 months.
Concentrations of Alpha 1 Anti Trypsin (AAT) levels in stool | From enrollment to the end of treatment at 3 months
  Alpha 1 Anti Trypsin (AAT) levels in stool samples were examined using ELISA (mcg/g). The differences in the concentrations of AAT levels between placebo and Inbumin Forte groups will be analysed after 3 months of treatment.
Concentrations of amino acid in blood samples | From enrollment to the end of treatment at 3 months
  Amino acids levels (µmol/l) in blood samples were examined using LC-MSMS. The differences of amino acid levels between placebo and Inbumin Forte will be analysed at the end of 3 months
Complete hematological profiles | From enrollment to the end of treatment at 3 months
  Complete hematological profiles in blood samples were examined using sysmex analyzer. The differences between placebo and Inbumin will be analysed at the end of 3 months.Time Frame: From enrollment to the end of treatment at 3 months
Iron status levels | From enrollment to the end of treatment at 3 months
  serum ferritin (ng/ml) were examined using mini vidas immunology analyzer, serum iron (µg/dL), total iron binding capacity (µg/dL) were examined using Vitros Chemistry analyzer. The differences between placebo and Inbumin will be analysed at the end of 3 months.Time Frame: From enrollment to the end of treatment at 3 months
Intestinal microbiota profiles | From enrollment to the end of treatment at 3 months
  Intestinal microbiota were examined using PCR technique. The differences between placebo and Inbumin will be analysed at the end of 3 months.Time Frame: From enrollment to the end of treatment at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Taniawati Supali, Study Chair — Indonesia University
Locations (2):
- Indonesia (2):
  - Indonesian territories, South Bangka Or Toboali, Bangka–Belitung Islands
  - IMERI Faculty of Medicine Universitas Indonesia, Central Jakarta, DKI Jakarta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Snakehead Fish (Channa striata) and Its Biochemical Properties for Therapeutics and Health Benefits
- [Background] Potential effect of Striatin (DLBS0333), a bioactive protein fraction isolated from Channa striata for wound treatment
- [Background] Lisowska-Myjak B, Pachecka J, Sokrates O, Brzozowska-Binda A, Torbicka E. Fecal alpha-1-antitrypsin excretion in children with diarrhea. Scand J Gastroenterol. 1998 Mar;33(3):255-9. doi: 10.1080/00365529850170829. PMID 9548618
- [Background] Li F, Ma J, Geng S, Wang J, Liu J, Zhang J, Sheng X. Fecal calprotectin concentrations in healthy children aged 1-18 months. PLoS One. 2015 Mar 5;10(3):e0119574. doi: 10.1371/journal.pone.0119574. eCollection 2015. PMID 25742018
- [Background] Vaz Nery S, Bennett I, Clarke NE, Lin A, Rahman Z, Rahman M, Clements ACA. Characterisation of environmental enteropathy biomarkers and associated risk factors in children in the context of a WASH trial in Timor-Leste. Int J Hyg Environ Health. 2018 Jul;221(6):901-906. doi: 10.1016/j.ijheh.2018.05.012. Epub 2018 Jun 8. PMID 29891218
- [Background] Semba RD, Shardell M, Sakr Ashour FA, Moaddel R, Trehan I, Maleta KM, Ordiz MI, Kraemer K, Khadeer MA, Ferrucci L, Manary MJ. Child Stunting is Associated with Low Circulating Essential Amino Acids. EBioMedicine. 2016 Apr;6:246-252. doi: 10.1016/j.ebiom.2016.02.030. Epub 2016 Feb 19. PMID 27211567
- [Background] Endrinikapoulos A, Afifah DN, Mexitalia M, Andoyo R, Hatimah I, Nuryanto N. Study of the importance of protein needs for catch-up growth in Indonesian stunted children: a narrative review. SAGE Open Med. 2023 Apr 17;11:20503121231165562. doi: 10.1177/20503121231165562. eCollection 2023. PMID 37101818
- [Background] Mrimi EC, Palmeirim MS, Minja EG, Long KZ, Keiser J. Malnutrition, anemia, micronutrient deficiency and parasitic infections among schoolchildren in rural Tanzania. PLoS Negl Trop Dis. 2022 Mar 4;16(3):e0010261. doi: 10.1371/journal.pntd.0010261. eCollection 2022 Mar. PMID 35245314
- [Background] Lahav-Ariel L, Caspi M, Nadar-Ponniah PT, Zelikson N, Hofmann I, Hanson KK, Franke WW, Sklan EH, Avraham KB, Rosin-Arbesfeld R. Striatin is a novel modulator of cell adhesion. FASEB J. 2019 Apr;33(4):4729-4740. doi: 10.1096/fj.201801882R. Epub 2018 Dec 28. PMID 30592649
- See also: Related Info — https://scienceforecastoa.com/Articles/SJBBE-V1-E1-1005.pdf
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/9548618/
- See also: Related Info — https://journals.plos.org/plosone/article?id=10.1371/journal.pone.0119574
- See also: Related Info — https://pmc.ncbi.nlm.nih.gov/articles/PMC4856740/
- See also: Related Info — https://pmc.ncbi.nlm.nih.gov/articles/PMC10123915/pdf/10.1177_20503121231165562.pdf
- See also: Related Info — https://pmc.ncbi.nlm.nih.gov/articles/PMC8926280/pdf/pntd.0010261.pdf
- See also: Related Info — https://pmc.ncbi.nlm.nih.gov/articles/PMC6988865/